CLINICAL TRIAL: NCT05349318
Title: Hyperbaric Oxygen Therapy for Prodromal Alzheimer´s Disease With Cerebrovascular Disease: A Prospective, Randomized, Double Blind Study
Brief Title: Hyperbaric Oxygen Therapy for Prodromal Alzheimer´s Disease With Cerebrovascular Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 254-21-ASF
Record Dates: First submitted 2022-03-21; First posted 2022-04-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Prodromal Alzheimer's Disease; Cerebral Vascular Disorder; Mild Cognitive Impairment; Vascular Cognitive Impairment
MeSH Terms: conditions — Cerebrovascular Disorders; Cognitive Dysfunction | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Upon consent and evaluation, eligible participants will be randomized with equal probability into one of two arms: HBOT or SHAM. The evaluation procedure will be performed at baseline, after the treatment and after a maintenance period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible candidates will be randomized with equal probability to the HBOT and sham interventions. Randomization will be performed using a computer software based on patients' code.
  Since the HBOT chamber can hold six subjects, the randomization will be done in clusters of six patients. After randomization, when a cluster of six subjects from one of the arms will be filled, the intervention for that cluster will begin.
  Three study technicians will be the only unblinded staff who have the key for the group assignment of each subject. They will exclusively activate the HBOT/sham protocol during session times. All subjects and other clinic staff will remain blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric Oxygen Therapy active arm (Active Comparator): The protocol comprises of 60 consecutive hyperbaric oxygen treatment (HBOT) sessions, 5 sessions per week within a three months' period. Then there will be a maintenance period for 6 months in which the participants will receive HBOT twice a week.
  Interventions: Device: Hyperbaric oxygen therapy
- Sham active arm (Sham Comparator): The protocol comprises of 60 consecutive Sham sessions, 5 sessions per week within a three months' period. Then there will be a maintenance period for 6 months in which the participants will receive Shan sessions twice a week.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — Each session will include exposure of 90 minutes to 100% at 2 ATA, with 5 minutes air breaks every 20 minutes
  Arms: Hyperbaric Oxygen Therapy active arm
Device: Sham — Each session will include exposure of 90 minutes to 21% at 1.2 ATA during the first five minutes of the session with the noise of circulating air, and then decrease slowly during the next five minutes to 1.03 ATA
  Arms: Sham active arm

SUMMARY:
Alzheimer´s disease is a devastating illness that effects the patients as well as their family members. Its prevalence increases exponentially and the burden on the healthcare system is enormous. AD neuropathology begins 15-20 years before the occurrence of cognitive symptoms, which ranges from preclinical stage to mild cognitive impairment (MCI) to dementia. Prodromal AD is an early stage of the disease which is characterized by positive biomarkers and MCI. To this day, there is no medication that can cure or halt the progression of the disease and most studies focus on finding reversible risk factors and changing their influence. Several aetiologies have been proposed, like the deposition of amyloid and tau proteins, neuroinflammation and cerebral ischemia due to cerebrovascular factors. The Amyloid deposition, which serves as the biological marker of AD, was originally thought to be the main cause of the disease, however, recent data suggests that it is not the cause and that it might actually has a protective role. On the other hand, it is known today that vascular changes with related tissue ischemia and neuroinflammation have a crucial role in the development of AD in many patients. These pathologies, ischemia & neuroinflammation, can be improved by the use of hyperbaric oxygen therapy (HBOT). The goal of this study is to explore the potential beneficial effect of HBOT on prodromal AD.

DETAILED DESCRIPTION:
Alzheimer disease is characterised by cognitive, mental and functional disability that is expected to progress until the patient is fully dependent on others for activities of daily living. The pathology begins many years until the cognitive symptoms appear. Prodromal Alzheimer's disease is a state where a person has mild cognitive impairment and Amyloid deposition, which is seen on brain Amyloid PET or in lumbar puncture.

To date, there has been neither a cure nor a therapy that can significantly halt or relieve symptoms for most patients.

This study offers a new biological therapeutic approach aimed to induce neuroplasticity and improve neurological and cognitive functions. Pre -clinical as well as clinical data indicate that HBOT can be beneficial for those patients who suffer from MCI due to Alzheimer's disease and also to patients with cerebral vascular disease.

HBOT is a well-known treatment used in clinical practice for other indications and is considered to be safe with relative rare mild and reversible side effect .The study is designed as a prospective, randomized, sham controlled double blinded study.

Subjects will be enrolled up to a total of 100 subjects, age 60-85, diagnosed with MCI and positive Amyloid PET and vascular changes on brain MRI.

Eligible patients will be randomized to the two study groups at a ratio of 6:6 (in clusters of 6 patients). The HBOT/sham treatment includes 60 daily sessions of 90 minutes each, five days per week. After the treatment period, there will be a maintenance period of HBOT/sham sessions twice a week for 6 months. All assessments with be done on baseline, after the treatment period and after the maintenance period.

The primary endpoint includes improvement in cognitive scores in neurocognitive evaluations (Neurotrax). Secondary and tertiary endpoints include changes in cognitive, physiological, physical, imaging, lab tests and self report questionaires.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Mild cognitive impairment (MCI) due to AD or mixed AD and vascular dementia pathology
2. MMSE score of 20 and above
3. Stable psychological and pharmacological treatment for more than three months prior to inclusion.
4. Caregiver that is seeing the patient at least twice per week and is willing to participate and accompany the patient and fill questionnaires
5. Subject willing and able to read, understand and sign an informed consent

Exclusion Criteria:

1. Inability to attend scheduled clinic visits and/or comply with the study protocol
2. History of traumatic brain injury, brain tumors, brain surgery, chronic subdural haemorrhages, Epilepsy
3. Active malignancy
4. Substance use at baseline, except for prescribed cannabis if vaporized or taken PO as tincture
5. History of other neurodegenerative diseases including Parkinson's disease (PD), Lewy body dementia (LBD), Frontotemporal dementia (FTD), Multiple sclerosis (MS), Amyotrophic lateral sclerosis (ALS), Creutzfeld Jacob disease (CJD), Multisystem atrophy (MSA), Pseudobulbar palsy (PSP), Corticobasal degeneration (CBD), Wernicke Korsakoff syndrome
6. Chronic use of medications that may compromise cognitive function and cannot be stopped: Anticonvulsants, Anticholinergics, antiparkinsonian, corticosteroids, Benzodiazepines
7. Moderate to severe sleep apnea with no use of CPAP
8. Diagnosis of a psychiatric disorder including: major depression, schizophrenia, bipolar disorder
9. Serious suicidal ideation
10. Renal or liver insufficiency, electrolyte imbalances
11. Chronic heart failure with ejection fraction of 35 or less
12. HBOT for any reason prior to study enrolment
13. Chest pathology incompatible with pressure changes (including active asthma or COPD)
14. Ear or Sinus pathology incompatible with pressure changes (above 3 otolaryngologist visits a year)
15. An inability to perform an awake brain MRI or Amyloid PET
16. An inability to perform computerized cognitive tests (Neurotrax)
17. MMSE score below 20
18. No evidence of amyloid in the brain PET
19. No evidence of vascular related lesions in the brain MRI
20. Active smoking
21. Participation in another study

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of neurocognitive functions evaluation by Mindstreams cognitive battery test (Neurotrax) | At baseline, 3 months
  Memory, attention and information process will be evaluated using the NeuroTrax computerized cognitive evaluation battery.
Change from baseline of neurocognitive functions evaluation by Mindstreams cognitive battery test (Neurotrax) | 9 months
  Memory, attention and information process will be evaluated using the NeuroTrax computerized cognitive evaluation battery.

SECONDARY OUTCOMES:
Brain amyloid PET using Flumetamol (Vizamyl) tracer | At baseline, 3 months, 9 months
  Brain amyloid assessment using PET scan with Flumetamol (Vizamyl) tracer will be used to assess change in amyloid burden
Whole-brain quantitative perfusion imaging | At baseline, 3 months, 9 months
  Whole-brain quantitative perfusion imaging will be performed using Dynamic susceptibility contrast (DSC)-MRI technique
Brain microstructure MRI evaluation | At baseline, 3 months, 9 months
  Fractional anisotropy (FA) and Mean diffusivity (MD) will be evaluated using diffusion tensor imaging (DTI) MRI protocol
Brain volume MRI evaluation | At baseline, 3 months, 9 months
  Gray matter and hippocampal volumetric measurement using high-resolution MP-RAGE 3D MRI
Brain functional connectivity imaging | At baseline ,3 months, 9 months
  Resting state functional MRI

OTHER OUTCOMES:
Quality of life SF-36 questionnaire | At baseline, 3 months, 9 months
  Self reported SF-36 quality of life questionnaire
The Pittsburgh Sleep Quality Index (PSQI) questionnaire | At baseline, 3 months, 9 months
  Self reported quality of sleep questionnaire
The Depression, Anxiety and Stress Scale-21 (DASS-21) | At baseline, 3 months, 9 months
  Self reported questionnaire of depression, anxiety and stress
Advanced Activities of Daily Function (a-ADL) | At baseline, 3 months, 9 months
  Questionnaire of activities of daily living for the patient and the informant
Clinical Dementia Rating (CDR) scale - sum of boxes | At baseline, 3 months, 9 months
  Cognitive assessment of 6 cognitive and functional domains, based on an interview of the patient and a reliable informant
Montreal Cognitive Assessment (MOCA) | At baseline, 3 months, 9 months
  Neurocognitive assessment
Mini Mental State Exam (MMSE) | At baseline, 3 months, 9 months
  Neurocognitive assessment
Serum inflammatory markers | At baseline, 3 months, 9 months
  Serum inflammatory markers include: IL-1, IL-6, tumor necrosis factor-alpha, hsCRP
Alzheimer's disease (AD) biomarkers: Abeta 42/40 | At baseline, 3 months, 9 months
  Plasma will be tested for Abeta 42/40
Alzheimer's disease (AD) biomarkers: P-tau181 | At baseline, 3 months, 9 months
  Plasma will be tested for P-tau181
Alzheimer's disease (AD) biomarkers: P-tau231 | At baseline, 3 months, 9 months
  Plasma will be tested for P-tau 231
Alzheimer's disease (AD) biomarkers: neurofilament light (NfL) | At baseline, 3 months, 9 months
  Plasma will be tested for neurofilament light (NfL)
Alzheimer's disease (AD) biomarkers: plasma glial fibrillary acidic protein (GFAP) | At baseline, 3 months, 9 months
  Plasma will be tested for plasma glial fibrillary acidic protein (GFAP)
Vascular biomarker- Vascular endothelial growth factor (VEGF) | At baseline, 3 months, 9 months
  Serum will be tested for VEGF
Passive behavioral monitoring using BHQ smartphone application | Through study completion, up to one year
  An application will be installed on the participants' smartphones for continuous passive monitoring of human behavior
Cardiopulmonary exercise test (CPET) | At baseline, 3 months, 9 months
  CPET determines the anaerobic threshold that is expected to change through the intervention
Neuro-physical evaluation - Static balance | At baseline, 3 months, 9 months
  Static balance will be assessed by the Balance Error Scoring System (BESS)
Neuro-physical evaluation- Timed Up and Go test | At baseline, 3 months, 9 months
  Dynamic balance and risk of falling will be assessed by the Timed Up and Go test (TUG)
Neuro-physical evaluation - 10 meter walk | At baseline, 3 months, 9 months
  Dynamic balance and risk of falling will be assessed by 10-meter walk (10MW).
Neuro-physical evaluation - Sit to Stand test | At baseline, 3 months, 9 months
  Muscle function will be assessed by the sit to stand (STS) test for the leg strength and endurance
Neuro-physical evaluation - Hand held dynamometery | At baseline, 3 months, 9 months
  Muscle function will be assessed by the hand-held dynamometry (HHD) for the isometric grip strength.
Neuro-physical evaluation - 6 minute walk | At baseline, 3 months, 9 months
  The sub-maximal aerobic capacity and endurance will be assessed by the 6-minute walk test (6MWT).
Event-related synchronization (ERS) change - EEG | At baseline, 3 months, 9 months
  The EEG will include a three-level visual N-back task, and go-no-go task
Event-related desynchronization (ERD) change - EEG | At baseline, 3 months, 9 months
  The EEG will include a three-level visual N-back task, and go-no-go task
Grand average P300 ERP change - EEG | At baseline, 3 months, 9 months
  The EEG will include a three-level visual N-back task, and go-no-go task
Alpha band power change - EEG | At baseline, 3 months, 9 months
  The EEG will include a three-level visual N-back task, and go-no-go task
Beta band power change - EEG | At baseline, 3 months, 9 months
  The EEG will include a three-level visual N-back task, and go-no-go task
Gamma band power change - EEG | At baseline, 3 months, 9 months
  The EEG will include a three-level visual N-back task, and go-no-go task
Delta band power change - EEG | At baseline, 3 months, 9 months
  The EEG will include a three-level visual N-back task, and go-no-go task
Theta to alpha bands power ratio change - EEG | At baseline, 3 months, 9 months
  The EEG will include a three-level visual N-back task, and go-no-go task
N-back match/no match percentage change - EEG | At baseline, 3 months, 9 months
  The EEG will include a three-level visual N-back task, and go-no-go task

CONTACTS AND LOCATIONS:
Overall Officials: Karin Elman Shina, MD, Principal Investigator — Senior Neurologist and director of the neuropsychology and physiology unit
Locations (1):
- Shamir Medical Center (Assaf Harofeh), Ẕerifin, Israel